CLINICAL TRIAL: NCT03104764
Title: Evaluation of Wound Healing and Patients´Experiences of Labial Frenulum Surgery - a Randomized, Controlled Comparative Study of Conventional Scalpel Technique and Er-Yag Laser Technique
Brief Title: Labial Frenulum Surgery - a Comparative Study of Conventional Scalpel and Er-Yag Laser Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Dental Health in Uppsala Region (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2014/253
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2014-09

CONDITIONS: Labial Tie
Keywords: labial frenulum; surgery; scalpel technique; Er:YAG laser
MeSH Terms: interventions — Laser Therapy; Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, single-blind investigation
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor have not met the patient before assessing the outcome. The assessor has no information about which surgical technique that is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalpel (Active Comparator): Frenotomy performed with conventional scalpel
  Interventions: Device: Scalpel
- Er:YAG laser (Experimental): Frenotomy performed with Er:YAG laser
  Interventions: Device: Er:YAG laser

INTERVENTIONS:
Device: Scalpel — Labial frenulum removed by scalpel
  Arms: Scalpel
Device: Er:YAG laser — Labial frenulum removed by Er:YAG laser
  Arms: Er:YAG laser

SUMMARY:
The aim of the study was to compare the outcome in terms of wound healing time, surgery time, bleeding and patient experience of the ectomy of frenulum when performed with laser technology versus conventional scalpel technique. A prospective, single-blind, randomized and controlled study was performed. Wound healing was assessed five and ten days after after surgery. The long-term outcome were assessed blinded by a dentist not earlier involved in the study.

DETAILED DESCRIPTION:
Children referred to a pediatric clinic to surgically remove a labial frenulum were randomized to treatment with conventional scalpel or laser treatment technology after parents and children had given consent to participate. During the surgery the time required for the procedure and the amount of bleeding the different techniques caused were measured. Wound healing was assessed five and ten days after surgery by a clinical judgement and by analysing photos. Three months after surgery an independent dentist assessed the long-term outcome by a clinical examination. The patients´ view of the treatment were assessed directly after the surgery and five days, ten days and three months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients in need of frenulum labials surgery

Exclusion Criteria:

* patients with severe general diseases (ASA>2)
* patients who required general anaesthesia for treatment

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-11-04 (Actual); Study Completion 2016-01-25 (Actual)

PRIMARY OUTCOMES:
Wound healing | 0-3 months
  Time period until reepithelialized measured clinically and on photos

SECONDARY OUTCOMES:
Patient experience | 0-3 months
  Patients´experiences of surgery procedures measured through questionnaires
Time required for surgery | Intervention day
  The time required for the surgical process is measured with timer
Scar tissue formation | 3 months
  prevalence of scar tissue formation assessed by a clinical investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Public Dental Service, Vretgränd 9, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not planned to be shared